CLINICAL TRIAL: NCT00004454
Title: Phase I/II Study of Retroviral-Mediated Transfer of Iduronate-2-Sulfatase Gene Into Lymphocytes of Patients With Mucopolysaccharidosis II (Mild Hunter Syndrome)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: University of Minnesota (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/13577; UMN-HUNTER; UMN-5P01HD32652
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-10

CONDITIONS: Mucopolysaccharidosis II
Keywords: inborn errors of metabolism; mucopolysaccharidosis; mucopolysaccharidosis II; rare disease
MeSH Terms: conditions — Mucopolysaccharidosis II; Metabolism, Inborn Errors; Mucopolysaccharidoses; Rare Diseases

INTERVENTIONS:
Genetic: lymphocyte gene therapy

SUMMARY:
OBJECTIVES: I. Evaluate the safety and feasibility of treating mucopolysaccharidosis II (mild Hunter syndrome) by lymphocyte gene therapy.

II. Determine the levels of iduronate-2-sulfatase enzyme in these patients attained by infusing increasing doses of lymphocytes transduced with a retroviral vector designed for insertion and expression of this iduronate-2-sulfatase gene (L2SN).

III. Determine the duration of survival of these transduced cells in these patients.

IV. Determine whether monthly infusion of L2SN-transduced lymphocytes accomplishes metabolic correction (as measured by glycosaminoglycan excretion), decrease in liver or spleen volume, any therapeutic effect upon cardiac and pulmonary dysfunction, or any other effects from treatment.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Peripheral blood lymphocytes are harvested from patient by apheresis, stimulated to initiate the growth of T-lymphocytes, transduced with retrovirus L2SN containing iduronate-2-sulfatase, and reinfused into the patient.

Patients receive 12 monthly infusions of these retroviral-mediated gene transduced lymphocytes with the first three infusions in a dose escalation format.

Patients are monitored for at least 2 hours after completion of each infusion. Patients are followed at 1 year after treatment, and then until death.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Mucopolysaccharidosis II (mild Hunter syndrome) as defined by the following:

* Characteristic coarse facial features, hepatosplenomegaly, and radiographic evidence of dysostosis multiplex
* Elevated urinary excretion of glycosaminoglycans in 3 urine specimens
* Deficient iduronate-2-sulfatase enzyme activity as measured in plasma and leukocytes
* Mutation consistent with mild Hunter syndrome must have either: A single base substitution of the coding sequence not previously associated with severe Hunter syndrome phenotype OR An exon-skipping mutation that would allow for occasional production of (minimal amounts of) normal protein

--Patient Characteristics--

Cardiovascular: No severe cardiac disease

Pulmonary: No severe respiratory disease

Other:

* Must have IQ score of 80 or higher
* Effective contraception required of all fertile patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2
Dates: Start 1996-10

CONTACTS AND LOCATIONS:
Overall Officials: Chester B. Whitley, Study Chair — University of Minnesota
Locations (1):
- University of Minnesota Medical School, Minneapolis, Minnesota, United States